CLINICAL TRIAL: NCT03343171
Title: Continuum™ Ceramic Bearing System in Total Hip Arthroplasty. A Multi-center, Prospective, Non-controlled Post Market Surveillance Study
Brief Title: Continuum Ceramic on Ceramic Bearing Post Market Clinical Follow-Up Study
Status: Active, not recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: 09-H02
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Osteoarthritis; Avascular Necrosis; Inflammatory Arthritis; Post-traumatic Arthritis
Keywords: total hip arthroplasty
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis; Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | US Export: Yes

SUMMARY:
The primary objective of this study is to obtain implant survivorship and clinical outcome data for the commercially available Zimmer® Continuum™ Ceramic-on-Ceramic Bearing System when used in primary hip arthroplasty. This will be done by analysis of standard scoring systems, radiographs and adverse event records. Data will be used to monitor pain, mobility and survivorship, and to confirm the safety and efficacy of the Continuum Ceramic-on-Ceramic Bearing System.

DETAILED DESCRIPTION:
The subject of this clinical investigation is the Continuum Ceramic Bearing THA System in primary total hip arthroplasty. This system consists of a cementless modular Trabecular Metal™ (TM) Continuum Acetabular Shell, a modular BIOLOX delta Taper liner, and a modular BIOLOX delta femoral head. The characteristics of this THA system may allow for reduction in wear and osteolysis as compared to other approved and marketed THA systems and thus increase the expected implant life. The study design will be a prospective, multicenter, non-comparative post-market study, involving orthopedic surgeons skilled in hip arthroplasty procedures. A total of 200 patients will be enrolled into the study distributed between 6 study centres. This number of clinical centers will permit assessment of consistency among a multitude of investigators. Follow-up visits will. be performed at 6 weeks, 6 months, 1,2, 3, 5; 7 and 10 years post-operatively. All potential study subjects will be required to participate in the Informed Consent Process.

The safety and performance of the Implant System will be assessed as following: implant survivorship based on revision with removal of the study device; safety based on incidence and frequency of adverse events; and Performance will be determined by comparing the overall pain and functional performances, survivorship, subject quality-of-life and radiographic parameters of study subjects who received the Continuum Ceramic Bearing System.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 21 to 75 years of age, inclusive.
* Patient is skeletally mature.
* Patient qualifies for primary unilateral or bilateral total hip arthroplasty (THA) based on physical exam and medical history including the following:

  * Avascular necrosis (AVN)
  * Osteoarthritis (OA)
  * Inflammatory arthritis (i.e. Rheumatoid arthritis)
  * Post-traumatic arthritis
* Patient has no history of previous prosthetic replacement device (any type, including surface replacement arthroplasty, endoprosthesis, etc.) of the affected hip joint(s).
* Patient has a Harris Hip Score <70 in the affected hip
* Patient is willing and able to provide written informed consent.
* Patient is willing and able to cooperate in the required post-operative therapy.
* Patient is willing and able to complete scheduled follow-up evaluations as described in the Informed Consent.
* Patient has participated in the Informed Consent process and has signed the Ethics Committee approved informed consent.

Exclusion Criteria:

* The patient is:

  * A prisoner
  * Mentally incompetent or unable to understand what participation in the study entails
  * A known alcohol or drug abuser
  * Anticipated to be non-compliant.
* The patient has a neuromuscular disorder, vascular disorder or other conditions that could contribute to prosthesis instability, prosthesis fixation failure, or complications in postoperative care.
* The patient has a vascular (large and small vessel disease) insufficiency.
* The patient has a chronic renal impairment or failure.
* The patient has had previous prosthetic hip replacement device (any type, including surface replacement arthroplasty, endoprosthesis, etc.) in the joint to be operated
* The patient has a neurologic condition in the ipsolateral or contralateral limb which affects lower limb function.
* The patient has a diagnosed systemic disease that could affect his/her safety or the study outcome.
* The patient is known to be pregnant.
* The patient is unwilling or unable to give informed consent, or to comply with the follow-up program.
* The patient has received an investigational drug or device within the previous 6 months.
* The patient has undergone a total hip replacement, endoprosthesis, or surface arthroplasty of the contralateral (opposite side) hip within the past 6 months regardless of whether the previous hip was enrolled in this clinical study.
* The patient has an active or latent infection in or about the affected hip joint or an infection distant from the hip joint that may spread to the hip hematogenously.
* The patient has had previous girdlestone procedure (resection arthroplasty) or surgical fusion of the hip to be operated.
* The patient has insufficient bone stock to fix the component. Insufficient bone stock exists in the presence of metabolic bone disease (i.e. osteoporosis), cancer, and radiation. Note: Dual Energy X-ray Absorptiometry (DEXA) may be used to assess the presence of adequate bone stock.
* The patient has known local bone tumors and/or cysts in the operative hip.
* The patient has a known sensitivity or allergic reaction to one or more of the implanted materials.
* The patient is Grade III obese with a Body Mass Index (BMI) > 35.
* The patient has osteoradionecrosis in the affected hip joint

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, suffering from severe hip pain and disability requiring total hip arthroplasty, who meet the inclusion/exclusion criteria and who receives the Continuum™ Ceramic Bearing System.
Sampling Method: Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2010-09-15 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Safety will be evaluated by adverse events reporting. | 10 years
  Safety will be evaluated by monitoring the frequency and incidence of adverse events (AE), serious adverse events (SAE), adverse device effects (ADE) and serious adverse device effects (SADE)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Achakri, Study Director — Zimmer Biomet
Locations (6):
- HYKS-instituutti Oy, Helsinki, Finland
- Italy (2):
  - Dipartimento di Ricerca Traslazionale e delle Nuove Tecnologie in Medicina e Chirurgia, Università di Pisa, Pisa
  - Policlinico Tor Vergata, Rome
- United Kingdom (3):
  - Glasgow Royal Infirmary, Glasgow
  - Nuffield Department of Orthopaedics, University of Oxford, Oxford
  - Southampton General Hospital, Southampton